CLINICAL TRIAL: NCT01183728
Title: Regeneration of Articular Cartilage in Grade II, III and IV Knee Osteoarthritis by Intraarticular Injection of Autologous Bone Marrow Stem Cells Expanded ex Vivo With a GMP Procedure Developed by IBGM-Valladolid (MSV)
Brief Title: Treatment of Knee Osteoarthritis With Autologous Mesenchymal Stem Cells
Acronym: KDD&MSV
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Red de Terapia Celular (Industry)
Collaborators: Fundacion Teknon, Centro Medico Teknon, Barcelona (Unknown); University of Valladolid (Other); Centro en Red de Medicina Regenerativa de Castilla y Leon (Other); Institut de Terapia Regenerativa Tissular (Other); EGARSAT Suma Intermutual, Barcelona, Spain (Unknown); Cetir Sant Jordi, S.a.. (Individual)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TerCel001; Eudra-CT 2009-017405-11 (Other Grant/Funding Number: RD06/0010/0000); Protocol Code (Registry Identifier: MSV-arthro-2009-01)
Record Dates: First submitted 2010-08-13; First posted 2010-08-18 (Estimated); Results first posted 2015-01-15 (Estimated); Last update posted 2015-01-15 (Estimated); Status verified 2015-01

CONDITIONS: Osteoarthritis, Knee; Knee Degenerative Disease; Knee Osteoarthritis
Keywords: Knee degenerative disease; osteoarthritis; gonarthrosis; stem cell; cellular therapy; regenerative therapy; Mesenchymal stem cells; Bone marrow; musculoskeletal Diseases
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis; Musculoskeletal Diseases | interventions — Genes, mos

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- MSV autologous transplantation (Experimental): Bone marrow collected from patient will be used for mesenchymal stem cells isolation and expansion under GMP conditions at IBGM-Valladolid (MSV). Autologous MSV implanted in knee by articular injection
  Interventions: Other: Autologous bone marrow mesenchymal stem cells (MSV)

INTERVENTIONS:
Other: Autologous bone marrow mesenchymal stem cells (MSV) — Bone marrow collection from patient, mesenchymal cells isolation and expansion under GMP conditions following the IBGM-Valladolid protocol (MSV). Autologous MSV implantation by articular injection.
  Other Names: MSV, mesenchymal stem cells by IBGM-Valladolid protocol.

SUMMARY:
In this prospective study we aim to evaluate the feasibility and safety of the implantation of 40 millions MSV in knees with osteoarthritis of grade II-IV (Kellgren and Lawrence). The working hypothesis proposes that MSV antiinflammatory effect will help healing of articular cartilage degeneration to a grade enough to be objectivized by questionnaires and imaging procedures. The study of quantitative changes in structure and composition of cartilage determined by MRI T2-mapping (Cartigram ) will be performed at 6, 12 and 24 months. Pain and disability will be assessed by visual analogue scale (VAS), WOMAC, Lequesne Index and evaluation of the quality of life by Short Form 36 questionnaire (SF-36) completed at 3, 6,12 and 24 months.

DETAILED DESCRIPTION:
Knee osteoarthritis is the most common form of arthritis. Treatments involve high costs in terms of social and economic, are palliative and do not contemplate healing by regenerative therapy. It has been shown recently, that mesenchymal stem cells (MSC) can be expanded "in vitro" and may regenerate several damaged or injured tissues. In addition its has demonstrated that MSC are able to modulate immune responses and to control inflammation through its action on T lymphocytes. Preliminary studies in animal models, including one carried out in an equine by our research group, confirms feasibility, safety and efficacy evidence proposed treatment protocol. Our research group has also experience in preparing clinical-grade MSC from bone marrow for other clinical trials and has all the necessary facilities and permissions to comply with GMPs imposed by recent EU legislation. Finally, our clinical team has a wide experience in regenerative therapies in several previous clinical trials for bone and cartilage.

We present here an alternative proposal, aiming to anti-inflammation and regeneration by injection of single dose of mesenchymal stem cells expanded from autologous bone marrow by the GMP-complying IBGM-Valladolid procedure (MSV). Treatment involves two non-invasive surgical procedures with low morbidity: obtaining bone marrow under local anesthesia and sedation, and 4 weeks later, articular injection of the cell product (20 millions MSVs). The injection of cells does not even require anesthesia and obtaining bone marrow requires an outpatient admission two hours following safety criteria.

Patients will be evaluated clinically, including pain score (VSA), pain and disability indexes (WOMAC and Lequesne) and life quality (SF-36), and by radiologic and MRI procedures no contrast and allowing quantification of morphological and structural changes of the cartilage region studied (MRI T2-mapping).

The design of the study is an open-label prospective, multicenter study. It will recruit 12 patients with osteoarthritis of II-IV Kellgren and Lawrence grades, Patients will be evaluated clinically by previous studies imaging (X-rays and MRI). If they are eligible for the study we shall provide them information about the clinical trial with the "Patient Information Sheet, quoting them for the Inclusion Visit. In the "Inclusion Visit" if the patient decides to participate in the test should sign the Informed Consent Document and a schedule for MRI and X-rays will be scheduled. The results of this exploration will be considered the standard to which compare any given change in the controls at 6 and 12 months. On this visit, routine preoperative examinations are performed (EKG, chest X-ray AP, basic analytic coagulation tests and identification of HIV, Lues and hepatitis B and C and the valuation by the Internal Medicine Service).

During the visit V0 we shall verify that all inclusion criteria persist and not exclusion criteria have appeared, and we shall program V1 (to obtain bone marrow) and provide a preliminary date for MSV injection 4 week later (V2). After application, the patients will have follow-up schedule at 8 days (V3), 3 (V4), 6 (V5), 12 (V6) and eventually 24 months (V7) as detailed below.

V0: Eligibility. Clinical History. Analysis, Imaging test. Programming of the following visits V1 (day 0): Bone marrow aspiration under local anesthesia and sedation V2 (day 23). MSV Implantation. V3 (+8 days from Implantation): Security evaluation. V4 (+3 months from Implantation): Security evaluation. VAS, WOMAC, Lequesne Index, SF-36 questionnaires.

V5 (+6 months from Implantation): Security evaluation. VAS, WOMAC, Lequesne Index, SF-36 questionnaires, RX, RNM.

V6 (+12 months from Implantation): Security evaluation. VAS, WOMAC, Lequesne Index, SF-36 questionnaires, RX, RNM.

V7 (+24 months from Implantation): Security evaluation. VAS, WOMAC, Lequesne Index, SF-36 questionnaires, RX, RNM.

ELIGIBILITY:
Inclusion Criteria:

* Knee osteoarthritis grade II, III and IV of Kellgren and Lawrence assessed by two observers.
* Chronic knee pain with mechanical characteristics.
* No local or systemic septic process.
* Haematological and biochemical analysis without significant alterations that contraindicate treatment.
* Informed written consent of the patient.
* The patient is able to understand the nature of the study

Exclusion Criteria:

* Age over 75 or under 18 years or legally dependent
* Any sign of infection
* Positive serology for HIV-1 or HIV-2, Hepatitis B (HBsAg, Anti-HCV-Ab), Hepatitis C (Anti-HCV-Ab) and syphilis.
* Congenital or acquired malformation resulting in significant deformity of the knee and leading to problems in application or evaluation of results.
* Overweight expressed as body mass index (BMI) greater than 30.5 (obesity grade II). BMI estimated as mass (kg) / corporal surface (m2).
* Women who are pregnant or intend to become pregnant or breast-feeding
* Neoplasia
* Immunosuppressive states
* Participation in another clinical trial or treatment with a different investigational product within 30 days prior to inclusion in the study.
* Other pathologic conditions or circumstances that difficult participation in the study according to medical criteria

Ages: 18 Years to 76 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2010-05; Primary Completion 2014-08 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Luis Orozco, MD, PhD, Principal Investigator — Fundacion Teknon; Ana Sanchez, MD, PhD, Study Director — IBGM, University of Valladolid; Robert Soler, MD, Study Director — Institut de Teràpia Regenerativa Tissular, Centro Médico Teknon; Javier Garcia-Sancho, MD, PhD, Study Director — IBGM, University of Valladolid
Locations (2):
- Spain (2):
  - Teknon Medical Center, ITRT, Barcelona, Barcelona
  - Instituto de Biologia y Genetica Molecular (IBGM), University of Valladolid, Valladolid, Valladolid

REFERENCES:
- [Result] Orozco L, Munar A, Soler R, Alberca M, Soler F, Huguet M, Sentis J, Sanchez A, Garcia-Sancho J. Treatment of knee osteoarthritis with autologous mesenchymal stem cells: a pilot study. Transplantation. 2013 Jun 27;95(12):1535-41. doi: 10.1097/TP.0b013e318291a2da. PMID 23680930
- [Result] Orozco L, Munar A, Soler R, Alberca M, Soler F, Huguet M, Sentis J, Sanchez A, Garcia-Sancho J. Treatment of knee osteoarthritis with autologous mesenchymal stem cells: two-year follow-up results. Transplantation. 2014 Jun 15;97(11):e66-8. doi: 10.1097/TP.0000000000000167. No abstract available. PMID 24887752
- See also: Spanish Cell Therapy Network — http://red-tercel.com
- See also: Cell application, ITRT-Centro Médico Teknon — http://www.itrt.es
- See also: Cell production, Instituto de Biologia y Genetica Molecular (IBGM) University of Valladolid — http://www.ibgm.med.uva.es
- See also: osteoarthritis, knee — http://www.ncbi.nlm.nih.gov/mesh/68010003

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | MSV Autologous Transplantation
Started | 12
Completed | 12
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: All included patients met the inclusion criteria and no exclusion criteria.
Arm/Group | MSV Autologous Transplantation
Number analyzed (Participants) | 12
Age, Customized [Number; unit: participants]
  >=18 and <=70 years | 9
  >70 years | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 8
Region of Enrollment [Number; unit: participants]
  Spain | 12
Number of Participants with Major Surgical History on Treated Knee [Number; unit: participants]
  With Major Surgical History on Treated Knee | 9
  Without Major Surgical History on Treated Knee | 3
Number of Participants with 4th grade osteoarthritis. [Number; unit: participants]
  With 4th grade osteoarthritis | 5
  With 2nd or 3th grade osteoarthritis | 7

OUTCOME MEASURES:

1. Primary Outcome: Feasibility and Safety of the Implementation of MSV in the Treatment of Osteoarthritis of the Knee.
Description: Clinical review, questionaires (VAS - Visual Analogue Scale (a psychometric response scale which can be used for subjective measurements of knee pain), WOMAC - Western Ontario and McMaster Universities Osteoarthritis Index (questionnaire to quantify the pain, stiffness and physical function in patients with osteoarthritis of the knee or hip), Lequesne Index (is a composite measure of pain and disability, with specific self-report questionnaires for knee (osteoarthritis)), SF36 life quality - Short Form 36 (is a questionnaire for the detection of changes in quality of life)).
  In all cases, the scale was from 0 to 100%. Measurements were performed before cell transplantation (0) and 3, 6, 12 and 24 months afterwards depending on the questionnaire. For VAS, WOMAC and Lequesne, lower values represent a better outcome. For SF-36, higher values represent a better outcome.
  VAS-DA, VAS for pain associated to daily activities. VAS-SP, VAS for pain associated to sports activities.
Time Frame: 0, 3, 6, 12 and 24 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | MSV Autologous Transplantation
Number analyzed (Participants) | 12
units on a scale
  Knee pain VAS-DA. 0 months | 46.9 (7.5)
  Knee pain VAS-DA. 3 months | 25.1 (6.8)
  Knee pain VAS-DA. 6 months | 24.8 (6.0)
  Knee pain VAS-DA. 12 months | 15.4 (3.8)
  Knee pain VAS-DA. 24 months | 15.8 (12.0)
  Knee pain VAS-SP. 0 months | 56.1 (5.1)
  Knee pain VAS-SP. 3 months | 29.8 (7.3)
  Knee pain VAS-SP. 6 months | 28.9 (6.4)
  Knee pain VAS-SP. 12 months | 18.5 (3.9)
  Knee pain VAS-SP. 24 months | 18.9 (5.3)
  WOMAC - Pain. 0 months | 24.2 (4.1)
  WOMAC - Pain. 12 months | 5.8 (1.6)
  WOMAC - Pain. 24 months | 11.7 (4.0)
  WOMAC - Rigidity. 0 months | 10.4 (3.7)
  WOMAC - Rigidity. 12 months | 5.2 (3.2)
  WOMAC - Rigidity. 24 months | 8.3 (4.2)
  WOMAC - Function loss. 0 months | 19.1 (3.8)
  WOMAC - Function loss. 12 months | 9.4 (3.2)
  WOMAC - Function loss. 24 months | 12.1 (6.1)
  WOMAC - Total. 0 months | 19.4 (3.6)
  WOMAC - Total. 12 months | 8.3 (2.7)
  WOMAC - Total. 24 months | 11.7 (5.4)
  Lequesne. 0 months | 45.1 (5.6)
  Lequesne. 12 months | 14.9 (4.1)
  Lequesne. 24 months | 13.9 (4.7)
  SF-36. Physical Function. Basal | 18.8 (22.9)
  SF-36. Physical Function. 3 months | 21.0 (27.3)
  SF-36. Physical Function. 6 months | 25.7 (28.4)
  SF-36. Physical Function. 12 months | 25.1 (22.4)
  SF-36. Physical Role. Basal | 31.1 (24.5)
  SF-36. Physical Role. 3 months | 36.9 (26.5)
  SF-36. Physical Role. 6 months | 38.6 (26.3)
  SF-36. Physical Role. 12 months | 47.7 (13.7)
  SF-36. Bodily Pain. Basal | 27.2 (19.6)
  SF-36. Bodily Pain. 3 months | 25.7 (17.8)
  SF-36. Bodily Pain. 6 months | 31.8 (22.1)
  SF-36. Bodily Pain. 12 months | 36.3 (23.8)
  SF-36. General Health. Basal | 64.8 (16.8)
  SF-36. General Health. 3 months | 58.5 (17.5)
  SF-36. General Health. 6 months | 65.2 (22.5)
  SF-36. General Health. 12 months | 63.3 (20.9)
  SF-36. Vitality. Basal | 58.3 (23.3)
  SF-36. Vitality. 3 months | 53.9 (26.1)
  SF-36. Vitality. 6 months | 56.8 (18.2)
  SF-36. Vitality. 12 months | 47.7 (13.7)
  SF-36. Social Function. Basal | 48.8 (22.7)
  SF-36. Social Function. 3 months | 47.3 (25.0)
  SF-36. Social Function. 6 months | 53.0 (24.8)
  SF-36. Social Function. 12 months | 44.2 (18.2)
  SF-36. Role Emotional. Basal | 54.2 (5.1)
  SF-36. Role Emotional. 3 months | 53.2 (4.0)
  SF-36. Role Emotional. 6 months | 53.2 (4.0)
  SF-36. Role Emotional. 12 months | 50.8 (9.0)
  SF-36. Mental Health. Basal | 68.1 (18.7)
  SF-36. Mental Health. 3 months | 61.0 (22.6)
  SF-36. Mental Health. 6 months | 61.8 (19.5)
  SF-36. Mental Health. 12 months | 63.3 (22.3)

2. Secondary Outcome: Indication of Efficacy
Description: Clinical exploration, questionaires (VAS, WOMAC, Lequesne Index, SF-36 life quality) at all the periods. To evaluate effectiveness through development of criteria for quantitative MRI (Cartigram) denoting regeneration of articular cartilage at 6, 12 and 24 months after the implantation of MSV.
  Magnetic Resonance imaging measurements of T2 relaxation (Cartigram) performed at 0, 6 and 12 months to quantify articular cartilage degeneration. The values (in milliseconds) are T1/2 for decay of the T2 MRI signals. Normal values are below 50 ms; values above 50 ms correspond to inflamed cartilage.
  Mean (SD) are expressed as the percent of values (of a total of 88 measurements) that are between 50 and 90 ms. A value =5 is considered normal (can be attained by chance). Values above 5 are considered pathological. The worst possible is 100.
Time Frame: 0, 6, 12, 24 months
Measure: Mean (Standard Deviation); unit: percentage of values
Arm/Group | MSV Autologous Transplantation
Number analyzed (Participants) | 12
percentage of values
  MRI T2 mapping. 0 months | 19.5 (7.9)
  MRI T2 mapping. 6 months | 15.4 (7)
  MRI T2 mapping. 12 months | 14.3 (6.3)
  MRI T2 mapping. 24 months | 13 (5.8)

ADVERSE EVENTS:
Time Frame: 24 months
Arm/Group | MSV Autologous Transplantation
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 11/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MSV Autologous Transplantation (N=12)
Post implantation pain (Musculoskeletal and connective tissue disorders) | 6 (8) — between days 1 and 6
Joint swelling (Musculoskeletal and connective tissue disorders) | 3 (3) — Attributable to overload
Unexpected inflammation with joint effusion (Musculoskeletal and connective tissue disorders) | 3 (3)
Contralateral knee pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Lumar pain (Musculoskeletal and connective tissue disorders) | 2 (4)
hamstring tendinitis (Musculoskeletal and connective tissue disorders) | 1 (1)
Contralateral knee surgery (Surgical and medical procedures) | 1 (1)
Dental implant (Surgical and medical procedures) | 1 (1)
Influenza (Infections and infestations) | 1 (1)
Gluten and lactose intolerance (Gastrointestinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes